CLINICAL TRIAL: NCT03529591
Title: Is the Reduction in Intraocular Pressure Achieved With Treatment of 180 Degrees Equivalent to Treatment of 360 Degrees With Selective Laser Trabeculoplasty (SLT)?
Brief Title: Is the Reduction in IOP After Treatment of 180 Degrees Equivalent to Treatment of 360 Degrees With SLT?
Acronym: SLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Tony Lin, Assistant Professor Ophthalmology, Western University, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111317
Record Dates: First submitted 2018-05-03; First posted 2018-05-18 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma of Both Eyes; Intraocular Pressure
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 180 deg selective laser trabeculoplasty (Active Comparator): The right eye of a patient is randomized to be treated with either 180 or 360 degrees selective laser trabeculoplasty (SLT). The fellow eye is treated with the opposite treatment, that is, if the right eye is treated with 180 degrees SLT, the left eye is treated with 360 degrees SLT. Intraocular pressure (IOP) response is assessed at 2 weeks, one, three and six months post treatment and compared to the alternative treatment arm, the fellow eye.
  Interventions: Device: Selective laser trabeculoplasty (SLT); Procedure: Selective laser trabeculoplasty
- 360 deg selective laser trabeculoplasty (Active Comparator): The right eye of a patient is randomized to be treated with either 180 or 360 degrees selective laser trabeculoplasty (SLT). The fellow eye is treated with the opposite treatment, that is, if the right eye is treated with 180 degrees SLT, the left eye is treated with 360 degrees SLT. Intraocular pressure (IOP) response is assessed at 2 weeks, one, three and six months post treatment and compared to the alternative treatment arm, the fellow eye.
  Interventions: Device: Selective laser trabeculoplasty (SLT); Procedure: Selective laser trabeculoplasty

INTERVENTIONS:
Device: Selective laser trabeculoplasty (SLT) — In this study, treatment naive patients with bilateral ocular hypertension or primary open angle glaucoma are treated with 180 degrees SLT in one eye and 360 degrees SLT in the contralateral eye. The primary outcome measure is assessing the response to SLT in both eyes and comparing the intraocular pressure outcomes between the two eyes of each patient.
  Other Names: Selective laser trabeculoplasty
Procedure: Selective laser trabeculoplasty — In this study, treatment naive patients with bilateral ocular hypertension or primary open angle glaucoma are treated with 180 degrees SLT in one eye and 360 degrees SLT in the contralateral eye. The primary outcome measure is assessing the response to SLT in both eyes and comparing the intraocular pressure outcomes between the two eyes of each patient.

SUMMARY:
The study is a prospective randomised controlled intervention comparing the intraocular pressure outcomes following Selective Laser Trabeculoplasty (SLT) treatment of 180 degrees SLT compared to 360 degrees in treatment naive patients with bilateral ocular hypertension or primary open angle glaucoma . The right eye of each patient will be randomised to receive either 180 or 360 degrees SLT, while the fellow eye will receive the opposite treatment. That is, if the right eye is randomised to 180 degrees SLT, then the left eye will receive 360 degrees SLT.

The primary objective is to assess the mean difference in intraocular pressure between two eyes of each participant. The mean difference in IOP will be assessed at two weeks and at one, three and six months after treatment with SLT.

Secondary outcomes include assessing whether there are differences in visual acuity, anterior chamber inflammation, visual field progression and the rate of complications between the two eyes treated with either 180° or 360° of selective laser trabeculoplasty. The complications assessed are those published in the literature including: pain, blurred vision, anterior chamber inflammation, IOP spike, and hyphaema. Additionally, participants will be given the opportunity to report symptoms experienced through free text.

DETAILED DESCRIPTION:
Potential patients will be identified by the Principal Investigator during a clinic visit. Pre-screening criteria is carried out by the co-investigator or the research co-ordinator. General eligibility criteria, inclusion and exclusion criteria are applied. The Research Co-ordinator approaches the patient and the SLT laser study is discussed with the patient. The patient is provided the Information Sheet and advised to contact the Research Coordinator if they wish to proceed. Informed consent is obtained if the patient wishes to proceed. Baseline data is collected and the right eye is randomised with the fellow eye to receive non randomised treatment.

SLT is performed in both eyes (180 degrees in 1 eye + 360 degrees in the fellow eye) during an office visit. IOP in both eyes is checked and recorded at one hour post treatment.

The patient returns for follow up at two weeks post SLT treatment visit. A complete ocular examination, including IOP, is undertaken. Complications and adverse events are assessed and recorded. Any change to eyedrops is recorded. Patients return at one, three and six months for review, and the same assessment as above is undertaken at each visit.

Enrolling is complete when 48 patients are enrolled. Patients are advised enrolling is complete.

Statistical analysis is undertaken to assess the mean change in IOP between the two treatments. Complications and adverse events are each treatment group are recorded. The study is submitted for publication and written communication is provided to each enrolled patient.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* IOP greater than 21mmHg (millimetres mercury)
* Glaucoma suspect
* Open angle glaucoma - primary or secondary
* Bilateral disease
* History of previous uncomplicated cataract surgery
* Willingness to be treated with selective laser trabeculoplasty
* Willingness to participate in the study, along with signed written consent

Exclusion Criteria:

* Age younger than 18 years
* Paediatric glaucoma
* Narrow or closed angles on gonioscopy
* History of ocular trauma
* Active or history of uveitis
* History of amblyopia
* History of, or, current steroid use - ocular, periocular or systemic
* History of any prior ocular laser - Argon laser trabeculoplasty (ALT), SLT or retinal laser
* Monocular patient
* Active proliferative diabetic retinopathy
* History of complicated cataract surgery
* Recent cataract surgery - within the last six months
* Unable to consent for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure response (physiological parameter) | Six months
  Is there a difference in the intraocular pressure response following SLT treatment of 180 degrees compared to SLT treatment of 360 degrees, in two eyes of the same patient treatment?

SECONDARY OUTCOMES:
The number of participants with treatment-related adverse events will be assessed by CTCAE v4.0. | Six months
  The adverse events/complications in eyes treated with 180 degrees SLT compared to 360 degrees SLT will be assessed and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lin, MD, Principal Investigator — Ivey Eye Institute, St Joseph's Healthcare, Western University, London, Ontario, Canada
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114